CLINICAL TRIAL: NCT00172731
Title: Measurement of Activity Participation for Persons With Schizophrenia Living in the Community
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: 9361701289; NSC93-2413-H002-015-SSS
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-12-21 (Estimated); Status verified 2005-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of the study is to develop a questionnaire on community occupational participation for persons with schizophrenia living in the community. In the International Classification of Functioning, Disability, and Health (ICF) recently revised by World Health Organization, activity participation is recognized as an important indication of health-related status. From the perspective of occupational therapy, the researcher intends to investigate the experiences of occupational participation among schizophrenic patients living in the community, and to develop a measuring tool for occupational participation accordingly.

The development of the Community Occupational Participation Questionnaire will be based on the result of a qualitative research project which the researcher is carrying out at the moment. The resultant questionnaire will provide a quantitative measure of community occupational participation for persons with schizophrenia, as well as a measurement tool of activity participation for health-related research studies. Furthermore, it may provide valuable information to the development of community psychiatric services.

This current study will take one year. Tasks to be accomplished include: building item pool, examining content validity of each item, pilot testing, item analysis, norm establishment, and testing reliability and validity. Data will be collected in different areas of Taiwan, and will be analyzed with the following methods: content validity ratio, item-total correlation, Cronbach's alpha, and confirmatory factor analysis. The study will result in an occupational participation questionnaire with norm, validity and reliability.

DETAILED DESCRIPTION:
First, the participants were informed the right and how to fill the self-report survey questionnare in. And then they began to complete the questionnare. After finishing it, the participants gave the questionnare back to the examinor and got a gift as a reward.

ELIGIBILITY:
Inclusion Criteria:

* person with Schizophrenia
* Must be able to read Chinese
* Majorly living in community

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-03; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Chinyu Wu, PhD, Study Chair — Department of Occupational Therapy, National Taiwan University
Locations (1):
- National Taiwan University, Taipei, Taiwan